CLINICAL TRIAL: NCT05888727
Title: Feasibility and Initial Efficacy of a Wheelchair Exercise-training Intervention for Persons With Multiple Sclerosis
Brief Title: Examining a Wheelchair Exercise-training Intervention for Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Illinois at Chicago (Other); Craig Hospital (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Stephanie Lee Silveira, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-SPH-23-0719; R03HD107615 (NIH)
Record Dates: First submitted 2023-05-05; First posted 2023-06-05 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training Intervention (Experimental)
  Interventions: Behavioral: Seated Physical activity INtervention for persons with MS, "SPIN" program- Intervention Condition
- Wellness Control (Active Comparator)
  Interventions: Behavioral: WEllness for Longevity Living with MS (WELL)- Control Condition

INTERVENTIONS:
Behavioral: Seated Physical activity INtervention for persons with MS, "SPIN" program- Intervention Condition — The proposed exercise training program is based on Social Cognitive Theory (SCT) for promoting aerobic and strength training in wheelchair users with MS. The 16-week program includes one-on-one video chats with a behavioral coach and various "tracks" for progressive increases in both strength and aerobic training. The proposed strength training includes 15 exercises with step-by-step instructions using resistance bands and/or wrist weights that were adapted for seated body-position that can be executed in a wheelchair. The proposed aerobic training is arm cycle ergometry; this is a low-cost and modifiable option that fits the needs of both power and manual wheelchair users. Other proposed equipment includes a comprehensive Training Manual, fitness tracker for use during exercise training sessions, and Rate of Perceived Exertion (RPE) scale for guiding individualized exercise intensity. The research team created 12 Newsletters that align with 12 proposed coaching calls.
  Arms: Exercise Training Intervention
Behavioral: WEllness for Longevity Living with MS (WELL)- Control Condition — The attention/contact wellness control condition will mirror the exercise training intervention condition, but focuses on implementing health behaviors other than physical activity (e.g., diet and emotional wellbeing). This program is an adapted version of the WellMS program from Prof. Motl's Phase III clinical trial (NCT03490240). The program is based on SCT principles of behavior change and integrates wellness resources from the National MS Society (NMSS). The research team has created 12 Newsletters that will be delivered on the same chat schedule as the exercise training intervention. All coaching chats and newsletters will occur with the same frequency as in the exercise training intervention condition. Participants will be provided with a participant manual, logbook, and calendar. Participants will work with their behavioral coach on goal setting specific to wellness behaviors.
  Arms: Wellness Control

SUMMARY:
The goal of this randomized controlled clinical trial is to examine the feasibility and initial efficacy of undertaking and delivering a novel, stakeholder-informed exercise training program for wheelchair users with multiple sclerosis. The main questions it aims to answer are:

* Is the study feasible as measured by participant recruitment (24 participants total), retention (80%), and safety (adverse events)?
* Is the study acceptable as measured by participant satisfaction and perceptions using an evaluation survey and semi-structured interviews?
* Is there significant change in following the 16-week study in metabolic health outcomes, MS symptoms, and exercise behavior change? Participants will be randomized to complete the 16-week SPIN exercise training program or WellMS attention/contact wellness program.

Researchers will compare the SPIN and WellMS groups to determine if there is a significant difference in metabolic health outcomes, MS symptoms, and exercise behavior change.

DETAILED DESCRIPTION:
The proposed study will use a randomized controlled design to examine the feasibility and initial efficacy of undertaking and delivering a novel, stakeholder-informed exercise training program for wheelchair users with MS compared with an attention/contact wellness control condition. Feasibility testing is essential for (a) learning if an intervention can be delivered and then (b) refining the approach before conducting an expensive, fully powered efficacy study. The primary outcome of interest is process and resource feasibility as measured by participant recruitment, retention, and safety. The secondary outcome of interest is acceptability, specifically participant satisfaction and perceptions, assessed through an evaluation survey and semi-structured interviews. The tertiary outcomes encompass scientific outcomes of interest for larger efficacy trials (i.e., metabolic health outcomes, MS symptoms, and exercise behavior change).

Twenty-four participants will be recruited and randomized to complete the 16-week SPIN exercise training program or WellMS attention/contact wellness program. Recruitment, screening, and enrollment will be completed by a graduate research assistant and the intervention will be delivered online by the PI through one-on-one behavioral coaching. Data regarding the primary, secondary, and tertiary outcomes will be collected at throughout the study period.

The proposed study includes three specific aims and hypotheses:

Specific Aim 1: Evaluate the feasibility (i.e., recruitment, retention, and safety) of an exercise training intervention and attention/contact wellness control condition delivered over a 16-week period in a sample of 24 adult wheelchair users with MS from the Dallas-Fort Worth Metroplex.

Hypothesis 1: The study protocol will be feasible in terms of reaching recruitment goals (n=24; 12 per group) within a one-year period, retaining 80% or more of those participants through the full 16-week study period, and safe in terms of <10% of participants reporting adverse events.

Specific Aim 2: Evaluate the acceptability (i.e., participant satisfaction and perceptions) of a 16-week exercise training intervention and attention/contact wellness control condition in a sample of 24 adult wheelchair users with MS from the Dallas-Fort Worth Metroplex.

Hypothesis 2: Participants in both conditions will report high satisfaction (mean rating 4/5 or greater) via formative evaluation surveys and positive perceptions regarding their assigned program via post-test interviews.

Specific Aim 3: Assess the scientific outcomes of interest (i.e., metabolic health, MS symptoms, and exercise behavior change) for determining effect size and sample size estimates in powering a future R01.

Hypothesis 3: The intervention exercise training program will lead to greater improvements in metabolic health outcomes (i.e., HbA1c, cholesterol, glucose, and triglycerides, MS symptoms (i.e., fatigue, pain, depression, and quality of life) and exercise behavior compared to the attention/control wellness program.

Procedures. All study procedures have been reviewed and approved by the University of North Texas Institutional Review Board. Interested participants will contact the graduate research assistant for a telephone screening, which includes a comprehensive description of the study followed by screening for inclusion criteria. Participants deemed eligible for the study will then be sent a consent form to review and sign using through DocuSign. When the graduate research assistant receives the signed consent form, participants will be mailed a pre-test/baseline assessment packet. The pre-test assessment packet will include Actigraph GT3X+ accelerometer and instructions to wear the accelerometer on the non-dominant wrist for 7 days as well as an order for blood sample collection at a Quest Diagnostics location that is convenient for them. Participants will complete a battery of questionnaires online using Qualtrics. When the graduate research assistant receives the accelerometer and notification that a blood sample has been collected, participants will be randomized using a random numbers sequence with concealed allocation (i.e., opaque sealed envelopes) by a member of the research team. Following randomization, participants will be mailed their condition-specific program materials as well as instructions for downloading Zoom. Participants will be provided an opportunity to complete technology training sessions prior to beginning the program to support individuals with limited digital literacy. Further, the research team will have 3 data-enabled devices for participants who lack hardware and/or Internet access. Post-test assessment of tertiary outcomes following the 16-week intervention will mirror baseline assessments. Participants will be asked to complete an additional evaluation questionnaire to assess satisfaction with the program and usability of intervention components. All participants will be invited to complete a post-test semi-structured interview via Zoom to provide feedback on their experiences and suggestions for refining the program. All participants will be compensated for completing each assessment, and an additional sum will be provided for those who complete the post-test interview.

Data Analyses. The analysis will use the intent-to-treat principle where participants will be analyzed in their randomization assignment. The focus of Specific Aims 1 & 2 is on feasibility of the study protocol. Descriptive statistics including frequencies and percentages will be used to assess Hypotheses 1 & 2. Hypothesis 2 is focused on equally favorable outcomes between conditions, which is important for guiding a future, larger efficacy study because if one condition is rated more favorably that would incorporate additional bias. If differences in feedback are identified, modifications to the appropriate condition will be made prior to fully-powered efficacy testing. The scientific outcomes in Hypothesis 3 (i.e., metabolic health outcomes, MS symptoms, and exercise behavior) will be examined using 2 time by 2 group mixed factor ANOVA with estimation of Cohen's d values for effect sizes. Participant's change in scientific outcomes will be further examined and compared with the >0.5 SD will be considered meaningful change based on benchmarks established in previous research.

Fidelity Monitoring. The research team is creating a fidelity monitoring protocol that aligns with the 5 domains outlined by the NIH Behavior Change Consortium adapted from a protocol led by the PI that was applied in a Phase-III clinical trial. The PI will serve as the behavioral coach given her experience as a behavioral coach in both physical activity and wellness conditions in 5 waves of the aforementioned clinical trial. The PI is not involved in outcome assessments and parallel scripts have been developed for each condition oriented toward the condition's content. The scripts include a check-in on the previous week, discussion of the week's Newsletter topic, and planning for the subsequent week. In line with our previous studies, randomly selected participant chats will be selected for fidelity monitoring to be completed; a Co-I will review the recorded session using a standard checklist to ensure systematic bias is not present.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of MS
* self-reported use of a wheelchair (i.e., manual wheelchair, power wheelchair, or scooter) >50% of the time
* age of 18 years or older
* relapse free for the past 30 days
* being non-active defined as not engaging in regular physical activity (30 minutes accumulated per day) on more than 2 days of the week during the previous 6 months (i.e., not meeting current physical activity guidelines for MS)

Exclusion Criteria:

* during telephone screening participants will complete an exercise pre-participation health screen and if participants report any symptoms or conditions contradictive of exercise then physician clearance will be required before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Silveira, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Silveira SL, Motl RW, Froehlich-Grobe K, Kay M. Feasibility, acceptability, and initial efficacy of a wheelchair exercise training program in persons with multiple sclerosis: study protocol for a parallel group randomized controlled trial. Disabil Rehabil Assist Technol. 2024 Nov;19(8):2998-3005. doi: 10.1080/17483107.2024.2332322. Epub 2024 Mar 22. PMID 38520055

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 24 participants enrolled, only 23 were randomized.
Period: Overall Study
Arm/Group | Exercise Training Intervention | Wellness Control
Started | 12 | 11
Completed | 10 | 10
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Training Intervention | Wellness Control | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.58 (12.94) | 61.18 (14.72) | 56.17 (14.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 6 | 8 | 14
  Black | 5 | 3 | 8
  Latino/a | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
Disease Duration [Mean (Standard Deviation); unit: years] | 10.91 (8.98) | 22.30 (12.05) | 15.7 (11.9)
Patient Determined Disease Steps [Median (Full Range); unit: score on a scale] — The PDDS is a patient-reported measure of disability in which participants select a score from 0 to 8, where 0 indicates normal function and 8 indicates being bedridden.
  score on a scale | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8]
Type of MS [Count of Participants; unit: Participants]
  Relapsing Remitting Multiple Sclerosis (RRMS) | 3 | 5 | 8
  Secondary Progressive Multiple Sclerosis (SPMS) | 1 | 3 | 4
  Primary Progressive Multiple Sclerosis (PPMS) | 8 | 3 | 11
Wheelchair type [Count of Participants; unit: Participants]
  Power wheelchair | 5 | 6 | 11
  Manual wheelchair | 5 | 1 | 6
  Power scooter | 2 | 4 | 6
Education [Count of Participants; unit: Participants]
  Less than College | 2 | 0 | 2
  1-3 Years of College | 4 | 3 | 7
  College Graduate or More | 6 | 8 | 14
Household Income [Count of Participants; unit: Participants]
  $50,000 or Less | 6 | 5 | 11
  $50,001 or Greater | 6 | 4 | 10
  Prefer to not respond | 0 | 2 | 2
Marital Status [Count of Participants; unit: Participants]
  Married | 5 | 6 | 11
  Single/Divorced/Separated/Widowed | 7 | 5 | 12
Employed [Count of Participants; unit: Participants]
  Yes | 2 | 2 | 4
  No | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Study Feasibility: Number of Participants Recruited
Description: Feasibility of the intervention will be measured based on reaching recruitment goals (n=24) within a one-year period.
Time Frame: 16-weeks
Measure: Count of Participants; unit: Participants
Groups:
- All Eligible Participants: All eligible participants
Arm/Group | All Eligible Participants
Number analyzed (Participants) | 24
Participants | 24

2. Primary Outcome: Study Feasibility: Number of Participants Retained
Description: Feasibility of the intervention will be measured based on retention of >80% of enrolled participants for the full 16-week study period.
Time Frame: 16-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise Training Intervention | Wellness Control
Number analyzed (Participants) | 12 | 11
Participants | 10 | 10

3. Primary Outcome: Study Feasibility: Number of Participants With Study-Related Adverse Events
Time Frame: 16-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise Training Intervention | Wellness Control
Number analyzed (Participants) | 12 | 11
Participants | 1 | 0

4. Secondary Outcome: Acceptability: Number of Participants With Positive Perceptions During Semi-Structured Interview
Description: Acceptability was assessed through semi-structured interviews conducted with participants. Positive perception was defined as participants expressing favorable views or satisfaction with the intervention. Reported is the number of participants who expressed positive perceptions during the interview.
Time Frame: 16-weeks
Population: Data were only collected from participants who completed a semi-structured interview.
Measure: Count of Participants; unit: Participants
Arm/Group | Exercise Training Intervention | Wellness Control
Number analyzed (Participants) | 9 | 8
Participants | 9 | 8

5. Secondary Outcome: Acceptability as Measured by the Post-intervention Acceptability Survey
Description: The post-intervention acceptability Survey total score ranges from 1 to 5, a higher score indicates greater acceptability.
Time Frame: 16-weeks
Population: Data was only collected from participants who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise Training Intervention | Wellness Control
Number analyzed (Participants) | 10 | 9
score on a scale | 4.5 (0.97) | 4.56 (0.53)

6. Other Pre Specified Outcome: Change of Physical Activity Levels Through the Godin Leisure-Time Exercise Questionnaire
Description: Physical activity will be assessed using the Godin Leisure-Time Exercise Questionnaire. Total Godin Leisure Time Exercise Questionnaire scores range from 0-119, with higher scores indicating more exercise behavior. Participants will complete this questionnaire at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Metabolic Health Outcomes: Triglycerides
Description: Triglycerides will be measured in partnership with Quest Diagnostics using the standard Diabetes Risk without Score panel at a location convenient to participants within their community. Participants will complete blood sample collection at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in Metabolic Health Outcomes: HbA1c
Description: HbA1c will be measured in partnership with Quest Diagnostics using the standard Diabetes Risk without Score panel at a location convenient to participants within their community. Participants will complete blood sample collection at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Change in Metabolic Health Outcomes: Cholesterol
Description: Cholesterol levels will be measured in partnership with Quest Diagnostics using the standard Diabetes Risk without Score panel at a location convenient to participants within their community. Participants will complete blood sample collection at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Change in Metabolic Health Outcomes: Glucose
Description: Fasting glucose will be measured in partnership with Quest Diagnostics using the standard Diabetes Risk without Score panel at a location convenient to participants within their community. Participants will complete blood sample collection at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Adherence to Assigned Condition
Description: We will ask all participants to complete a weekly form in an individual REDCap portal with the information from their logbook as an additional measure of adherence to the exercise training or wellness program (i.e., behavior change).
Time Frame: 16-weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in MS Symptoms: Fatigue
Description: Fatigue will be assessed using the Fatigue Severity Scale. Fatigue Severity Scale scores range from 9-63, with higher scores indicating greater fatigue. Participants will complete this questionnaire at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in MS Symptoms: Pain
Description: Pain will be assessed using the McGill Pain Questionnaire-Short Form. McGill Pain Questionnaire-Short Form scores range from 0-45, with higher scores indicating greater pain. Participants will complete this questionnaire at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in MS Symptoms: Depression
Description: Depressive symptoms will be assessed using the Hospital Anxiety and Depression Scale. Hospital Anxiety and Depression Scale depression subscale scores range from 0-21, with higher scores indicating greater depressive symptoms. Participants will complete this questionnaire at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Change in MS Symptoms: Quality of Life
Description: Quality of life will be assessed using the 12-item Short Form Survey. The 12-item Short Form Survey scores include mental and physical component subscale scores, which each range from 0-100, with higher scores indicating greater quality of life. Participants will complete this questionnaire at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Change of Physical Activity Levels Through Accelerometery From Baseline at 16 Weeks
Description: Physical activity will be assessed using an ActiGraph accelerometer. Participants will wear an accelerometer on a wristband on their nondominant wrist during the waking hours of a 7 day period. Participants will complete this at baseline and 16 weeks.
Time Frame: 16-weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 16 weeks
Arm/Group | Exercise Training Intervention | Wellness Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 4/12 | 2/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exercise Training Intervention (N=12) | Wellness Control (N=11)
Urinary tract infection (UTI) Hospitalization (Renal and urinary disorders) | 1 (1) | 0 (0)
Cognitive Hospital (Nervous system disorders) | 0 (0) | 1 (1)
Back Pain Cycling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
X-ray Slip Disk (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Minor MS Exacerbation (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT05888727/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-29): https://cdn.clinicaltrials.gov/large-docs/27/NCT05888727/ICF_001.pdf